CLINICAL TRIAL: NCT04390763
Title: A Phase II, Open Label, Randomized, Parallel Arm Study of NIS793 (With and Without Spartalizumab) in Combination With SOC Chemotherapy Gemcitabine/Nab-paclitaxel, and Gemcitabine/Nab-paclitaxel Alone in First-line Metastatic Pancreatic Ductal Adenocarcinoma (mPDAC)
Brief Title: Study of Efficacy and Safety of NIS793 (With and Without Spartalizumab) in Combination With SOC Chemotherapy in First-line Metastatic Pancreatic Ductal Adenocarcinoma (mPDAC)
Acronym: daNIS-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was early terminated following the NIS793 treatment halt and urgent safety measure issued in July 2023, as the continued evaluation of Standard of Care alone will not support the original purpose of this phase 2 clinical trial.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNIS793B12201; 2020-000349-14 (EudraCT Number)
Record Dates: First submitted 2020-05-14; First posted 2020-05-18 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Metastatic Pancreatic Ductal Adenocarcinoma
Keywords: NIS793; spartalizumab; gemcitabine; nab-paclitaxel; mPDAC; TGFβ; PD-1; Phase II
MeSH Terms: interventions — NIS-793; spartalizumab; Gemcitabine; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Safety Run-in (Experimental): Combination of NIS793 + spartalizumab + gemcitabine + nab-paclitaxel
  Interventions: Biological: NIS793; Biological: Spartalizumab; Drug: gemcitabine; Drug: nab-paclitaxel
- Randomized Arm 1 (Experimental): Combination of NIS793 + spartalizumab + gemcitabine + nab-paclitaxel
  Interventions: Biological: NIS793; Biological: Spartalizumab; Drug: gemcitabine; Drug: nab-paclitaxel
- Randomized Arm 2 (Experimental): Combination of NIS793 + gemcitabine + nab-paclitaxel
  Interventions: Biological: NIS793; Drug: gemcitabine; Drug: nab-paclitaxel
- Randomized Arm 3 (Active Comparator): gemcitabine + nab-paclitaxel
  Interventions: Drug: gemcitabine; Drug: nab-paclitaxel

INTERVENTIONS:
Biological: NIS793 — anti-TGFb antibody. NIS793 2100 mg every 2 weeks by intravenous (i.v.) infusion.
  Arms: Randomized Arm 1; Randomized Arm 2; Safety Run-in
Biological: Spartalizumab — anti-PD-1 antibody. spartalizumab 400 mg every 4 weeks by i.v. infusion.
  Other Names: PDR001
  Arms: Randomized Arm 1; Safety Run-in
Drug: gemcitabine — SOC chemotherapy. Gemcitabine (1000 mg/m^2 on Days 1, 8, and 15) i.v. given as per label.
Drug: nab-paclitaxel — SOC chemotherapy. Nab-paclitaxel (125 mg/m^2 on Days 1, 8, and 15) i.v. given as per label.
  Other Names: abraxane

SUMMARY:
The purpose of this Phase II study is to assess the efficacy and safety of NIS793 with and without spartalizumab in combination with gemcitabine/nab-paclitaxel versus gemcitabine/nab-paclitaxel in previously untreated mPDAC.

DETAILED DESCRIPTION:
This is a randomized, parallel arms, open-label, multi-center, Phase II study to evaluate the efficacy and safety of NIS793 with and without spartalizumab in combination with gemcitabine/nab-paclitaxel in participants with first-line metastatic pancreatic ductal adenocarcinoma (mPDAC).

The study started with a Safety Run-in to assess the safety and tolerability of NIS793 in combination with spartalizumab and standard of care (SOC) gemcitabine/nab-paclitaxel. Doses defined for each study treatment, as part of this quadruplet were administered in the Randomized part in the quadruplet/triplet/doublet-based treatment arms.

The Randomized part opened after the Safety Run-in had completed. Participants were randomized in a 1:1:1 ratio to one of the three treatment arms:

* Arm 1: NIS793 with spartalizumab and gemcitabine/nab-paclitaxel
* Arm 2: NIS793 with gemcitabine/nab-paclitaxel
* Arm 3: gemcitabine/nab-paclitaxel

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent must be obtained prior to participation in the study.
2. Male or female ≥ 18 years of age at the time of informed consent.
3. Participants with histologically or cytologically confirmed treatment-naïve metastatic adenocarcinoma of the pancreas with measurable disease as per RECIST 1.1.
4. Participants must have a site of disease amenable to biopsy, and be candidate for tumor biopsy according to the treating institution's guidelines. Participants must be willing to undergo a tumor biopsy at screening and during therapy on the study. In the event a new biopsy cannot be safely performed at study entry, an archival sample (collected <6 months prior) may be substituted following documented discussion with Novartis.
5. ECOG performance status ≤ 1.

Exclusion Criteria:

1. Previous radiotherapy, surgery (with exception of placement of biliary stent, which is allowed), chemotherapy or any other investigational therapy for the treatment of metastatic pancreatic cancer. Participants having received previous chemotherapy in the adjuvant setting.
2. Participants amenable to potentially curative resection.
3. Participants with a diagnosis of pancreatic neuroendocrine tumors (NETs), acinar, or islet cell tumors.
4. Having out of range laboratory values as pre-defined in the protocol.
5. Participants with MSI-H pancreatic adenocarcinoma.
6. Presence of symptomatic CNS metastases, or CNS metastases that require local CNS directed therapy (such as radiotherapy or surgery), or increasing doses of corticosteroids 2 weeks prior to study entry.
7. History of severe hypersensitivity reactions to any ingredient of study drug(s) and other mAbs and/or their excipients.
8. The participant exhibits any of the events outlined in the contra-indications or special warnings and precautions sections of gemcitabine and nab-paclitaxel as per locally approved labels.
9. Impaired cardiac function or clinically significant cardiac disease.
10. Known history of testing positive HIV infection.
11. Active HBV or HCV infection. Participants whose disease is controlled under antiviral therapy should not be excluded.
12. History of or current interstitial lung disease or pneumonitis grade ≥ 2
13. High risk of clinically significant gastrointestinal tract bleeding or any other condition associated with or history of significant bleeding.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-05-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (5):
  - Winship Cancer Institute, Atlanta, Georgia
  - Sidney Kimmel CCC At JH, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Cente, Boston, Massachusetts
  - Univ of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
- Australia (2):
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Liège, Belgium
- Novartis Investigative Site, Brno, Czech Republic, Czechia
- Novartis Investigative Site, Helsinki, Finland
- France (2):
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Toulouse
- Germany (3):
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Ulm
- Italy (3):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Verona, VR
- Novartis Investigative Site, Singapore, Singapore
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Sankt Gallen
  - Novartis Investigative Site, Zurich
- Taiwan (2):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2577

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 31 investigative sites in 14 countries.
Pre-assignment Details: The screening period began once patients had signed the study informed consent. Screening evaluations had to be completed within 21 days prior to the first dose of study treatment (≤ 28 days for baseline radiological assessments). After screening, the treatment period started on Cycle 1 Day 1.
Groups:
- Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel: NIS793 2100 mg every 2 weeks i.v. with spartalizumab 400 mg every 4 weeks i.v and standard of care chemotherapy in the safety run-in part
- Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel: NIS793 2100 mg every 2 weeks i.v. with spartalizumab 400 mg every 4 weeks i.v and standard of care chemotherapy in the randomized part
- Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel: NIS793 2100 mg every 2 weeks i.v. with standard of care chemotherapy in the randomized part
- Arm 3: Gemcitabine/Nab-paclitaxel: Standard of care chemotherapy in the randomized part
Period: Safety run-in Part
Arm/Group | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Started | 11 | 0 | 0 | 0
Safety Set 1 (All patients who received at least one dose of study treatment in the Safety run-in part.) | 11 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 11 | 0 | 0 | 0
Not completed — Adverse Event | 4 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Progressive Disease | 6 | 0 | 0 | 0
Period: Randomized Part
Arm/Group | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Started | 0 | 50 | 51 | 52
Full Analysis Set (FAS) (All patients to whom study treatment was assigned by randomization.) | 0 | 50 | 51 | 52
Safety Set 2 (All patients who received at least one dose of study treatment in the Randomized part.) | 0 | 46 | 49 | 45
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 50 | 51 | 52
Not completed — Adverse Event | 0 | 11 | 5 | 5
Not completed — Death | 0 | 3 | 4 | 2
Not completed — Physician Decision | 0 | 2 | 2 | 9
Not completed — Progressive Disease | 0 | 24 | 31 | 23
Not completed — Study terminated by sponsor | 0 | 1 | 0 | 0
Not completed — Participant Decision | 0 | 5 | 7 | 6
Not completed — Not treated | 0 | 4 | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel | Total
Number analyzed (Participants) | 11 | 50 | 51 | 52 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (8.77) | 64.3 (10.91) | 64.2 (9.90) | 64.8 (8.25) | 64.4 (9.59)
Age, Customized [Count of Participants; unit: Participants]
  18 - <65 years | 5 | 20 | 23 | 23 | 71
  65 - <85 years | 6 | 30 | 28 | 29 | 93
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 21 | 21 | 20 | 67
  Male | 6 | 29 | 30 | 32 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 39 | 35 | 33 | 116
  Black or African American | 0 | 1 | 1 | 3 | 5
  Asian | 2 | 9 | 15 | 15 | 41
  Unknown | 0 | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety run-in Part: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: A dose-limiting toxicity (DLT) is defined as an adverse event or abnormal laboratory value of Common Terminology Criteria for Adverse Events (CTCAE) grade ≥ 3 where the relationship to study treatment cannot be ruled out and is not clearly related solely to disease, disease progression, inter-current illness or concomitant medications, which occurs within the DLT evaluation period. The DLT evaluation period is the first 28 days of treatment with NIS793 with spartalizumab in combination with gemcitabine/nab-paclitaxel. Other clinically significant toxicities may be considered to be DLTs, even if not CTCAE grade 3 or higher.
Time Frame: First cycle of treatment (28 days)
Population: Dose-Determining Set (DDS) including all participants in the Safety run-in part who met the minimum exposure criterion defined in the protocol and had sufficient safety evaluations after 4 weeks of treatment or experienced a DLT during the first 4 weeks of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 6
Participants
  Any DLT | 1
  Colitis | 1

2. Primary Outcome: Safety run-in Part: Number of Participants With AEs and SAEs During the On-treatment Period
Description: Number of participants with AEs (any adverse events regardless of seriousness) and serious adverse events (SAEs), including changes from baseline in vital signs, electrocardiograms and laboratory results qualifying and reported as AEs.
  AE grades to characterize the severity of the AEs were based on the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. For CTCAE v5.0, Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening; Grade 5 = death related to AE.
  The on-treatment period is defined from the day of first administration of any study treatment up to 30 days after the date of the last actual administration of any study drug.
Time Frame: Up to approximately 0.8 years
Population: Safety set 1
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 11
Participants
  AEs | 11
  Treatment-related AEs | 11
  AEs with grade>=3 | 11
  Treatment-related AEs with grade>=3 | 8
  SAEs | 8
  Treatment-related SAEs | 3
  Fatal SAEs | 1
  Treatment-related fatal SAEs | 0

3. Primary Outcome: Safety run-in Part: Number of Participants With Dose Reductions and Dose Interruptions of NIS793, Spartalizumab, Gemcitabine and Nab-paclitaxel
Description: Number of participants with at least one dose reduction and at least one dose interruption of study drugs. Dose adjustments were permitted for patients who did not tolerate the protocol-specified dosing schedule.
  No dose reductions were allowed for NIS793 and spartalizumab beyond the first 28 days period of Safety run-in part.
Time Frame: Up to approximately 0.7 years
Population: Safety set 1
Measure: Count of Participants; unit: Participants
Arm/Group | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 11
Participants
  NIS793: At least one dose reduction or interruption | 5
  NIS793: At least one dose reduction | 0
  NIS793: At least one dose interruption | 5
  Spartalizumab: At least one dose reduction or interruption | 3
  Spartalizumab: At least one dose reduction | 0
  Spartalizumab: At least one dose interruption | 3
  Gemcitabine: At least one dose reduction or interruption | 9
  Gemcitabine: At least one dose reduction | 2
  Gemcitabine: At least one dose interruption | 9
  Nab-paclitaxel: At least one dose reduction or interruption | 9
  Nab-paclitaxel: At least one dose reduction | 3
  Nab-paclitaxel: At least one dose interruption | 9

4. Primary Outcome: Safety run-in Part: Dose Intensity of NIS793 and Spartalizumab
Description: Dose intensity of NIS973 and spartalizumab was calculated as cumulative actual dose in milligrams divided by duration of exposure in days and multiplied by 28 days. Dose adjustments were permitted for patients who did not tolerate the protocol-specified dosing schedule.
Time Frame: Cycle 1 and Cycle 3. The duration of each cycle was 28 days.
Population: Patients in the Safety set 1 who received NIS793 or spartalizumab at each reported treatment cycle.
Measure: Mean (Standard Deviation); unit: mg per cycle
Arm/Group | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 11
mg per cycle
  NIS793 - cycle 1 | 3627.3 (980.91)
  NIS793 - cycle 3: number analyzed (Participants) | 5
  NIS793 - cycle 3 | 4200.0 (0.00)
  Spartalizumab - cycle 1 | 400.0 (0.00)
  Spartalizumab - cycle 3: number analyzed (Participants) | 5
  Spartalizumab - cycle 3 | 400.0 (0.00)

5. Primary Outcome: Safety run-in Part: Dose Intensity of Gemcitabine and Nab-paclitaxel
Description: Dose intensity of gemcitabine and nab-paclitaxel was calculated as cumulative actual dose in milligrams/m^2 divided by duration of exposure in days and multiplied by 28 days.
Time Frame: Cycle 1 and Cycle 3. The duration of each cycle was 28 days.
Population: Patients in the Safety set 1 who received gemcitabine or nab-paclitaxel at each reported treatment cycle.
Measure: Mean (Standard Deviation); unit: mg per m^2 per cycle
Arm/Group | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 11
mg per m^2 per cycle
  Gemcitabine - cycle 1 | 2425.4 (698.27)
  Gemcitabine - cycle 3: number analyzed (Participants) | 5
  Gemcitabine - cycle 3 | 2619.1 (508.19)
  Nab-paclitaxel - cycle 1 | 303.3 (87.18)
  Nab-paclitaxel - cycle 3: number analyzed (Participants) | 5
  Nab-paclitaxel - cycle 3 | 327.6 (63.65)

6. Primary Outcome: Randomized Part: Progression-Free Survival (PFS) Per RECIST v1.1 - Bayesian Model
Description: PFS was based on local review of tumor assessments, using Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria. PFS is defined as the time from the date of randomization to the date of the first documented progression or death due to any cause. If a subject had not had an event, PFS was censored at the date of last adequate tumor assessment.
  PFS was estimated using a Bayesian model. For each comparison (arm 1 versus arm 3 and arm 2 versus arm 3), PFS was modeled using a two-piece hazard model, with specifying hazard rates before and after the possible delayed effect for arms 1 and 2 and constant hazard rate for arm 3.
  Results in the table as expressed as estimated posterior median hazard rate and one-sided 90% credible interval.
Time Frame: Up to approximately 2 years. Risk changing timepoint=approximately 0.3 years.
Population: Full Analysis Set (FAS)
Measure: Median (90% Confidence Interval); unit: events (progression, death) per year
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 50 | 51 | 52
events (progression, death) per year
  Hazard rate before the risk changing timepoint | 2.54 [0 to 3.34] | 1.23 [0 to 1.79] | 2.09 [0 to 2.53]
  Hazard rate after the risk changing timepoint | 1.46 [0 to 2.06] | 2.94 [0 to 3.86] | 2.09 [0 to 2.53]
Statistical Analysis 1: Comparison: Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel vs Arm 3: Gemcitabine/Nab-paclitaxel; Test type: Other; Bayesian two-piece hazard model; Hazard Ratio (HR) = 0.70, 90% CI 1-sided [upper limit 1.04] — Estimated posterior median of the HR after the risk changing timepoint and one-sided 90% credible interval are reported
Statistical Analysis 2: Comparison: Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel vs Arm 3: Gemcitabine/Nab-paclitaxel; Test type: Other; Bayesian two-piece hazard model; Hazard Ratio (HR) = 1.41, 90% CI 1-sided [upper limit 1.96] — Estimated posterior median of the HR after the risk changing timepoint and one-sided 90% credible interval are reported

7. Primary Outcome: Randomized Part: Progression-Free Survival (PFS) Per RECIST v1.1 - Kaplan-Meier Curves and Cox Model
Description: PFS was based on local review of tumor assessments, using RECIST 1.1 criteria. PFS is defined as the time from the date of randomization to the date of the first documented progression or death due to any cause. If a subject had not had an event, PFS was censored at the date of last adequate tumor assessment.
  PFS was analyzed based on the Kaplan-Meier curves and the Cox model.
Time Frame: Up to approximately 2 years
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 50 | 51 | 52
months | 3.91 [3.06 to 6.93] | 5.52 [3.94 to 7.29] | 4.37 [3.55 to 7.20]
Statistical Analysis 1: Comparison: Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel vs Arm 3: Gemcitabine/Nab-paclitaxel; Test type: Other; p = 0.46, Regression, Cox; Hazard Ratio (HR) = 1.02, 90% CI 1-sided [upper limit 1.37]
Statistical Analysis 2: Comparison: Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel vs Arm 3: Gemcitabine/Nab-paclitaxel; Test type: Other; p = 0.38, Regression, Cox; Hazard Ratio (HR) = 1.08, 90% CI 1-sided [upper limit 1.44]

8. Secondary Outcome: Randomized Part: Number of Participants With AEs and SAEs During the On-treatment Period
Description: as for outcome 2
Time Frame: Up to approximately 1.8 years
Population: Safety set 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 46 | 49 | 45
Participants
  AEs | 45 | 49 | 43
  Treatment-related AEs | 45 | 45 | 38
  AEs with grade>=3 | 42 | 42 | 35
  Treatment-related AEs with grade>=3 | 34 | 37 | 24
  SAEs | 32 | 26 | 26
  Treatment-related SAEs | 19 | 12 | 12
  Fatal SAEs | 3 | 1 | 4
  Treatment-related fatal SAEs | 1 | 0 | 0

9. Secondary Outcome: Randomized Part: Number of Participants With Dose Reductions and Dose Interruptions of NIS793, Spartalizumab, Gemcitabine and Nab-paclitaxel
Description: Number of participants with at least one dose reduction and at least one dose interruption of study drugs. Dose adjustments were permitted for patients who did not tolerate the protocol-specified dosing schedule.
  No dose reductions were allowed for NIS793 and spartalizumab in the Randomized part.
Time Frame: Up to approximately 1.7 years
Population: Safety set 2
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 46 | 49 | 45
Participants
  NIS793: At least one dose reduction or interruption: number analyzed (Participants) | 46 | 49 | 0
  NIS793: At least one dose reduction or interruption | 35 | 31 |
  NIS793: At least one dose reduction: number analyzed (Participants) | 46 | 49 | 0
  NIS793: At least one dose reduction | 0 | 0 |
  NIS793: At least one dose interruption: number analyzed (Participants) | 46 | 49 | 0
  NIS793: At least one dose interruption | 35 | 31 |
  Spartalizumab: At least one dose reduction or interruption: number analyzed (Participants) | 46 | 0 | 0
  Spartalizumab: At least one dose reduction or interruption | 21 |  |
  Spartalizumab: At least one dose reduction: number analyzed (Participants) | 46 | 0 | 0
  Spartalizumab: At least one dose reduction | 0 |  |
  Spartalizumab: At least one dose interruption: number analyzed (Participants) | 46 | 0 | 0
  Spartalizumab: At least one dose interruption | 21 |  |
  Gemcitabine: At least one dose reduction or interruption | 38 | 41 | 32
  Gemcitabine: At least one dose reduction | 25 | 23 | 19
  Gemcitabine: At least one dose interruption | 35 | 36 | 29
  Nab-paclitaxel: At least one dose reduction or interruption | 39 | 43 | 34
  Nab-paclitaxel: At least one dose reduction | 26 | 27 | 19
  Nab-paclitaxel: At least one dose interruption | 34 | 37 | 32

10. Secondary Outcome: Randomized Part: Dose Intensity of NIS973 and Spartalizumab
Description: as for outcome 4
Time Frame: Cycle 1 and Cycle 3. The duration of each cycle was 28 days
Population: Patients in the Safety set 2 who received NIS793 or spartalizumab at each reported treatment cycle.
Measure: Mean (Standard Deviation); unit: mg per cycle
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 46 | 49 | 0
mg per cycle
  NIS793 - cycle 1 | 3515.2 (995.32) | 3857.1 (784.22) |
  NIS793 - cycle 3: number analyzed (Participants) | 26 | 42 | 0
  NIS793 - cycle 3 | 3796.2 (844.03) | 3550.0 (982.59) |
  Spartalizumab - cycle 1: number analyzed (Participants) | 46 | 0 | 0
  Spartalizumab - cycle 1 | 400.0 (0.00) |  |
  Spartalizumab - cycle 3: number analyzed (Participants) | 24 | 0 | 0
  Spartalizumab - cycle 3 | 400.0 (0.00) |  |

11. Secondary Outcome: Randomized Part: Dose Intensity of Gemcitabine and Nab-paclitaxel
Description: as for outcome 5
Time Frame: Cycle 1 and Cycle 3. The duration of each cycle was 28 days
Population: Patients in the Safety set 2 who received gemcitabine or nab-paclitaxel at each reported treatment cycle
Measure: Mean (Standard Deviation); unit: mg per m^2 per cycle
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 46 | 49 | 45
mg per m^2 per cycle
  Gemcitabine - cycle 1 | 2442.3 (675.34) | 2644.8 (543.43) | 2392.1 (651.00)
  Gemcitabine - cycle 3: number analyzed (Participants) | 29 | 42 | 29
  Gemcitabine - cycle 3 | 2293.9 (710.08) | 2426.5 (696.10) | 2445.3 (561.36)
  Nab-paclitaxel - cycle 1 | 305.7 (84.91) | 330.7 (67.95) | 298.8 (80.96)
  Nab-paclitaxel - cycle 3: number analyzed (Participants) | 29 | 42 | 29
  Nab-paclitaxel - cycle 3 | 286.2 (86.45) | 296.2 (88.06) | 299.1 (70.08)

12. Secondary Outcome: Randomized Part: Overall Response Rate (ORR) Per RECIST v1.1
Description: ORR is the percentage of patients with a confirmed best overall response of complete response (CR) or partial response (PR), based on local investigator assessment per Response Evaluation Criteria for Solid Tumors (RECIST) v1.1.
  For RECIST v1.1, CR=Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR= At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Up to approximately 1.7 years
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 50 | 51 | 52
percentage of participants | 22.0 [11.5 to 36.0] | 31.4 [19.1 to 45.9] | 15.4 [6.9 to 28.1]

13. Secondary Outcome: Randomized Part: Duration of Response (DOR) Per RECIST v1.1
Description: DOR per RECIST v1.1 is defined as the time from the first documented response of CR or PR to the date of the first documented progression or death. DOR only applies to patients with a best overall response of CR or PR by investigator assessment per RECIST v1.1. Participants continuing without progression or death were censored at the date of their last adequate tumor assessment.
  DOR was analyzed using the Kaplan-Meier method.
Time Frame: Up to approximately 1.7 years
Population: Participants in the Full Analysis Set (FAS) with CR or PR
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 11 | 16 | 8
months | 7.75 [5.09 to NA] — Not estimable due to insufficient number of participants with events. | 4.86 [3.71 to 7.39] | 11.70 [3.61 to 16.20]

14. Secondary Outcome: Randomized Part: Time to Progression (TTP) Per RECIST v1.1
Description: TTP per RECIST v1.1 is defined as the time from the date of randomization to the date of event defined as the first documented progression per RECIST v1.1 or death due to underlying cancer. If a participant had no progression or death, the participant was censored at the date of last adequate tumor assessment.
  DOR was analyzed using the Kaplan-Meier method.
Time Frame: Up to approximately 1.7 years
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 50 | 51 | 52
months | 3.94 [3.55 to 7.03] | 5.59 [4.57 to 7.36] | 5.36 [3.68 to 8.61]

15. Secondary Outcome: Randomized Part: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of randomization to the date of death due to any cause.
  OS was analyzed using the Kaplan-Meier method.
Time Frame: Up to approximately 2 years
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 50 | 51 | 52
months | 10.7 [7.2 to 12.7] | 8.5 [7.7 to 9.9] | 10.1 [6.5 to 13.4]

16. Secondary Outcome: Randomized Part: Change From Baseline in PD-L1 Expression
Description: The tumor expression of programmed cell death-ligand 1 (PD-L1) was measured by immunohistochemical methods. Results are expressed as absolute change from baseline in PD-L1 expression.
Time Frame: Baseline (Screening), on-treatment (anytime between Cycle 3 Day 2 and Day 4). The duration of each cycle was 28 days.
Population: Participants in the Full Analysis Set (FAS) who had a valid assessment of PD-L1 tumor expression at both baseline and on-treatment.
Measure: Mean (Standard Deviation); unit: percentage of PD-L1 positive tumor cells
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 4 | 12 | 5
percentage of PD-L1 positive tumor cells | 7.625 (10.4193) | 7.917 (17.0572) | 4.000 (8.9443)

17. Secondary Outcome: Randomized Part: Change From Baseline in CD8 Expression
Description: The tumor expression of CD8 was measured by immunohistochemical methods. Results are expressed as absolute change from baseline in CD8 expression.
Time Frame: Baseline (Screening), on-treatment (anytime between Cycle 3 Day 2 and Day 4). The duration of each cycle was 28 days.
Population: Participants in the Full Analysis Set (FAS) who had a valid assessment of CD8 tumor expression at both baseline and on-treatment.
Measure: Mean (Standard Deviation); unit: percentage of CD8 marker area expression
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 3 | 14 | 6
percentage of CD8 marker area expression | 10.1 (11.01) | 1.4 (2.64) | 2.1 (1.82)

18. Secondary Outcome: Randomized Part: Number of Participants With Anti-NIS793 Antibodies
Description: The immunogenicity (IG) against NIS793 was assessed in serum using a validated enhanced electrochemiluminescence immunoassay (ECLIA).
  Patient anti-drug antibodies (ADA) status was defined as follows:
  * ADA-negative at baseline: ADA-negative sample at baseline
  * ADA-positive at baseline: ADA-positive sample at baseline
  * ADA-negative post-baseline: patient with ADA-negative sample at baseline and at least 1 post baseline sample, all of which are ADA-negative samples
  * ADA-inconclusive post-baseline = patient who does not qualify as ADA-positive or ADA-negative post-baseline
  * Treatment-induced ADA-positive = ADA-negative sample at baseline and at least 1 treatment-induced ADA-positive sample
Time Frame: Baseline (before first dose) and post-baseline (assessed throughout the treatment up to approximately 1.7 years)
Population: Participants in the safety set 2 who received NIS793 and had a non-missing baseline ADA sample and at least one non-missing post-baseline ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 41 | 44
Participants
  ADA-negative at baseline | 41 | 44
  ADA-positive at baseline | 0 | 0
  ADA-negative post-baseline | 41 | 44
  ADA- inconclusive post-baseline | 0 | 0
  Treatment-induced ADA-positive | 0 | 0

19. Secondary Outcome: Randomized Part: Number of Participants With Anti-spartalizumab Antibodies
Description: The immunogenicity (IG) against spartalizumab was assessed in serum using a validated a validated homogenous enzyme-linked immunosorbent assay (ELISA).
  Patient anti-drug antibodies (ADA) status was defined as follows:
  * ADA-negative at baseline: ADA-negative sample at baseline
  * ADA-inconclusive at baseline: patient who does not qualify as ADA-positive or ADA-negative at baseline
  * ADA-positive at baseline: ADA-positive sample at baseline
  * ADA-negative post-baseline: patient with ADA-negative sample at baseline and at least 1 post baseline sample, all of which are ADA-negative samples
  * ADA-inconclusive post-baseline = patient who does not qualify as ADA-positive or ADA-negative post-baseline
  * Treatment-induced ADA-positive = ADA-negative sample at baseline and at least 1 treatment-induced ADA-positive sample
Time Frame: Cycle 1 and Cycle 3. The duration of each cycle was 28 days
Population: Participants in the safety set 2 who received spartalizumab and had a non-missing baseline ADA sample and at least one non-missing post-baseline ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 41
Participants
  ADA-negative at baseline | 40
  ADA- inconclusive at baseline | 1
  ADA-positive at baseline | 0
  ADA-negative post-baseline | 35
  ADA- inconclusive post-baseline | 2
  Treatment-induced ADA-positive | 4

20. Secondary Outcome: Randomized Part: Maximum Observed Serum Concentration (Cmax) of NIS793
Description: Pharmacokinetic (PK) parameters were calculated based on NIS793 serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed concentration following a dose.
Time Frame: Cycle 1 and Cycle 3: pre-dose, 1, 24, 168 and 336 hours after the end of the infusion on Day 1. The duration of the infusion was 30 minutes. One cycle=28 days
Population: Participants in the pharmacokinetic analysis set (PAS) who received NIS793 and had an available value for the outcome measure. PAS consisted of all patients who received one dose (complete infusion) of the planned treatments and provided at least one valid primary PK parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 42 | 39
ng/mL
  Cycle 1 | 603000 (181000) | 622000 (192000)
  Cycle 3: number analyzed (Participants) | 21 | 31
  Cycle 3 | 821000 (235000) | 784000 (286000)

21. Secondary Outcome: Randomized Part: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of NIS793
Description: PK parameters were calculated based on NIS793 serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: as for outcome 20
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 42 | 39
h*ng/mL
  Cycle 1 | 84700000 (29300000) | 96000000 (26100000)
  Cycle 3: number analyzed (Participants) | 21 | 31
  Cycle 3 | 153000000 (52300000) | 151000000 (55000000)

22. Secondary Outcome: Randomized Part: Trough Serum Concentration (Ctrough) of NIS793
Description: Ctrough is defined as the concentration reached immediately before the next dose is administered. All drug concentrations below the lower limit of quantification were treated as zero for the calculation of PK parameters.
Time Frame: Cycle 1: pre-dose on Day 1. Cycle 3: pre-dose on Day 1 and Day 15 (combined). One cycle=28 days
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 26 | 34
ng/mL
  Cycle 1 | 137000 (51700) | 156000 (50100)
  Cycle 3: number analyzed (Participants) | 22 | 34
  Cycle 3 | 289000 (121000) | 291000 (126000)

23. Secondary Outcome: Randomized Part: Maximum Observed Serum Concentration (Cmax) of Spartalizumab
Description: PK parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed concentration following a dose.
Time Frame: Cycle 1 and Cycle 3: pre-dose, 1, 24, 168 and 648 hours after the end of the infusion on Day 1. The duration of the infusion was 30 minutes. One cycle=28 days
Population: Participants in the pharmacokinetic analysis set (PAS) who received spartalizumab and had an available value for the outcome measure. PAS consisted of all patients who received one dose (complete infusion) of the planned treatments and provided at least one valid primary PK parameter.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 42
µg/mL
  Cycle 1 | 109 (22.4)
  Cycle 3: number analyzed (Participants) | 21
  Cycle 3 | 120 (38.0)

24. Secondary Outcome: Randomized Part: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Spartalizumab
Description: PK parameters were calculated based on spartalizumab serum concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: as for outcome 23
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: h*µg/mL
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 42
h*µg/mL
  Cycle 1 | 10800 (4900)
  Cycle 3: number analyzed (Participants) | 21
  Cycle 3 | 3240 (1900)

25. Secondary Outcome: Randomized Part: Trough Serum Concentration (Ctrough) of Spartalizumab
Description: as for outcome 22
Time Frame: Cycle 2, 3 and 4: pre-dose on Day 1. One cycle=28 days
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 32
µg/mL
  Cycle 2 | 22.3 (8.67)
  Cycle 3: number analyzed (Participants) | 21
  Cycle 3 | 31.9 (11.7)
  Cycle 4: number analyzed (Participants) | 23
  Cycle 4 | 30.5 (14.3)

26. Secondary Outcome: Randomized Part: Maximum Observed Plasma Concentration (Cmax) of Gemcitabine
Description: PK parameters were calculated based on gemcitabine plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed concentration following a dose.
Time Frame: Cycle 1 and Cycle 4: pre-dose, end of infusion, and 2, 3, 5 and 24 hours after the start of infusion on Day 1. The duration of the infusion was according to the product labelling and local guidance. One cycle=28 days
Population: Participants in the pharmacokinetic analysis set (PAS) who received gemcitabine and had an available value for the outcome measure. PAS consisted of all patients who received one dose (complete infusion) of the planned treatments and provided at least one valid primary PK parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 42 | 40 | 44
ng/mL
  Cycle 1 | 9830 (8580) | 12000 (6850) | 10600 (6170)
  Cycle 4: number analyzed (Participants) | 23 | 28 | 24
  Cycle 4 | 7950 (5650) | 8830 (6150) | 7000 (4210)

27. Secondary Outcome: Randomized Part: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Gemcitabine
Description: PK parameters were calculated based on gemcitabine plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: as for outcome 26
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 42 | 40 | 44
h*ng/mL
  Cycle 1 | 7270 (6950) | 9900 (6140) | 8040 (4490)
  Cycle 4: number analyzed (Participants) | 23 | 28 | 24
  Cycle 4 | 5270 (4730) | 5980 (4410) | 4920 (2830)

28. Secondary Outcome: Randomized Part: Trough Serum Concentration (Ctrough) of Gemcitabine
Description: as for outcome 22
Time Frame: Cycle 4: pre-dose on Day 1. One cycle=28 days
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 24 | 30 | 23
ng/mL | 0 (0) | 0 (0) | 0 (0)

29. Secondary Outcome: Randomized Part: Maximum Observed Plasma Concentration (Cmax) of Nab-paclitaxel
Description: PK parameters were calculated based on nab-paclitaxel plasma concentrations by using non-compartmental methods. Cmax is defined as the maximum (peak) observed concentration following a dose.
Time Frame: as for outcome 26
Population: Participants in the pharmacokinetic analysis set (PAS) who received nab-paclitaxel and had an available value for the outcome measure. PAS consisted of all patients who received one dose (complete infusion) of the planned treatments and provided at least one valid primary PK parameter.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 37 | 38 | 43
ng/mL
  Cycle 1 | 9990 (37100) | 4120 (3370) | 3490 (1760)
  Cycle 4: number analyzed (Participants) | 19 | 28 | 24
  Cycle 4 | 4570 (4910) | 4050 (2410) | 2900 (1370)

30. Secondary Outcome: Randomized Part: Area Under the Serum Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUClast) of Nab-paclitaxel
Description: PK parameters were calculated based on nab-paclitaxel plasma concentrations by using non-compartmental methods. The linear trapezoidal method was used for AUClast calculation.
Time Frame: as for outcome 26
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 37 | 38 | 43
h*ng/mL
  Cycle 1 | 15700 (52400) | 5080 (2820) | 4820 (2500)
  Cycle 4: number analyzed (Participants) | 19 | 28 | 24
  Cycle 4 | 5960 (3650) | 5020 (3050) | 4250 (2550)

31. Secondary Outcome: Randomized Part: Trough Serum Concentration (Ctrough) of Nab-paclitaxel
Description: as for outcome 22
Time Frame: Cycle 4: pre-dose on Day 1. One cycle=28 days
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 19 | 30 | 23
ng/mL | 455 (1320) | 2.13 (10.4) | 3.25 (5.08)

32. Post Hoc Outcome: All-Collected Deaths
Description: On-treatment and post-treatment safety follow-up (FU) deaths were collected from first dose of study treatment to 90 days after last dose of NIS793, 150 days after last dose of spartalizumab and 30 days after last dose of gemcitabine and nab-paclitaxel, whichever was longer.
  Survival FU deaths were collected from 91 days after last dose of NIS793, 151 days after last dose of spartalizumab and 31 days after last dose of gemcitabine and nab-paclitaxel, whichever was longer, until end of study.
  All deaths refer to the sum of pre-treatment deaths, on-treatment and post-treatment safety FU deaths, and survival FU deaths.
Time Frame: On-treatment and post-treatment safety FU deaths: up to approximately 1 year (run-in part) and 1.9 years (randomized part). Survival FU deaths: up to approximately 1.8 years (run-in part) and 2 years (randomized part)
Population: Safety set 1 (safety run-in) and Full Analysis Set (randomized part)
Measure: Number; unit: Participants
Arm/Group | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel | Arm 3: Gemcitabine/Nab-paclitaxel
Number analyzed (Participants) | 11 | 50 | 51 | 52
Participants
  On-treatment and post-treatment safety FU deaths | 5 | 18 | 19 | 4
  Survival FU deaths: number analyzed (Participants) | 6 | 28 | 30 | 41
  Survival FU deaths | 5 | 15 | 22 | 35
  All deaths | 10 | 33 | 41 | 39

ADVERSE EVENTS:
Time Frame: On- and post-treatment safety FU: from first dose of study treatment to 90 days after last dose of NIS793, 150 days after last dose of spartalizumab and 30 days after last dose of gemcitabine and nab-paclitaxel, whichever was longer, up to approx. 1 year (run-in part) and 1.9 years (randomized part). Deaths in survival period: after completing safety FU until end of study, up to approx. 1.8 years (run-in part) and 2 years (randomized part).
Description: Deaths in the survival period are not considered Adverse Events (AEs). No AEs were collected in the survival period. Deaths were assessed in the Safety set 1 (run-in part) and Full Analysis Set (randomized part). AEs were assessed in the Safety set 1 (run-in part) and Safety set 2 (randomized part).
Groups:
- Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_On- and Post-treatment; Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_On- and Post-treatment; All Participants_On- and Post-treatment: Safety data up to 90 days after last dose of NIS793, 150 days after last dose of spartalizumab and 30 days after last dose of gemcitabine and nab-paclitaxel, whichever was longer
- Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel_On- and Post-treatment: Safety data up to 90 days after last dose of NIS793 and 30 days after last dose of gemcitabine and nab-paclitaxel, whichever was longer
- Arm 3: Gemcitabine/Nab-paclitaxel_On- and Post-treatment: Safety data up to 30 days after last dose of gemcitabine and nab-paclitaxel
- Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_Survival Period; Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_Survival Period: Deaths collected in the survival follow-up period (starting from Day 90 after last dose of NIS793, Day 151 days after last dose of spartalizumab and Day 31 after last dose of gemcitabine and nab-paclitaxel, whichever was longer). No AEs were collected during this period.
- Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel_Survival Period: Deaths collected in the survival follow-up period (starting from Day 90 after last dose of NIS793 and Day 31 after last dose of gemcitabine and nab-paclitaxel, whichever was longer). No AEs were collected during this period.
- Arm 3: Gemcitabine/Nab-paclitaxel_Survival Period: Deaths collected in the survival follow-up period (starting from Day 31 after last dose of gemcitabine and nab-paclitaxel). No AEs were collected during this period.
Arm/Group | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_On- and Post-treatment | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_On- and Post-treatment | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel_On- and Post-treatment | Arm 3: Gemcitabine/Nab-paclitaxel_On- and Post-treatment | All Participants_On- and Post-treatment | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_Survival Period | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_Survival Period | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel_Survival Period | Arm 3: Gemcitabine/Nab-paclitaxel_Survival Period
All-Cause Mortality (participants affected / at risk) | 5/11 | 18/50 | 19/51 | 4/52 | 46/164 | 5/6 | 15/28 | 22/30 | 35/41
Serious Adverse Events (participants affected / at risk) | 8/11 | 34/46 | 28/49 | 26/45 | 96/151 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 11/11 | 45/46 | 48/49 | 40/45 | 144/151 | 0/0 | 0/0 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_On- and Post-treatment (N=11) | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_On- and Post-treatment (N=46) | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel_On- and Post-treatment (N=49) | Arm 3: Gemcitabine/Nab-paclitaxel_On- and Post-treatment (N=45) | All Participants_On- and Post-treatment (N=151) | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_Survival Period (N=0) | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_Survival Period (N=0) | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel_Survival Period (N=0) | Arm 3: Gemcitabine/Nab-paclitaxel_Survival Period (N=0)
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 6 | 2 | 10 | NA | NA | NA | NA
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 1 | 4 | NA | NA | NA | NA
Haemolysis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Glucocorticoid deficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Hypopituitarism (Endocrine disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 3 | 6 | NA | NA | NA | NA
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Colitis (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 5 | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 0 | 5 | 0 | 0 | 5 | NA | NA | NA | NA
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Duodenal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Duodenal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Gastritis haemorrhagic (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | NA | NA | NA | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Ileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Impaired gastric emptying (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Melaena (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | NA | NA | NA | NA
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Subileus (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | NA | NA | NA | NA
Asthenia (General disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Chest pain (General disorders) | 0 | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Chills (General disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Fatigue (General disorders) | 0 | 3 | 0 | 0 | 3 | NA | NA | NA | NA
Gait inability (General disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Pain (General disorders) | 1 | 1 | 1 | 1 | 4 | NA | NA | NA | NA
Pyrexia (General disorders) | 2 | 5 | 3 | 5 | 15 | NA | NA | NA | NA
Biliary obstruction (Hepatobiliary disorders) | 0 | 1 | 2 | 0 | 3 | NA | NA | NA | NA
Cholangitis (Hepatobiliary disorders) | 0 | 2 | 2 | 0 | 4 | NA | NA | NA | NA
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Gallbladder rupture (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Abdominal infection (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | NA | NA | NA | NA
Acarodermatitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Biliary sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Biliary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 2 | NA | NA | NA | NA
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
COVID-19 pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Campylobacter infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Device related infection (Infections and infestations) | 0 | 0 | 3 | 0 | 3 | NA | NA | NA | NA
Febrile infection (Infections and infestations) | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA
Infection (Infections and infestations) | 0 | 3 | 1 | 0 | 4 | NA | NA | NA | NA
Large intestine infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 1 | 4 | 0 | 0 | 5 | NA | NA | NA | NA
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Pneumonia pseudomonal (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Postoperative wound infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Relapsing fever (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Sepsis (Infections and infestations) | 0 | 4 | 3 | 3 | 10 | NA | NA | NA | NA
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 2 | NA | NA | NA | NA
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0 | 2 | NA | NA | NA | NA
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
General physical condition abnormal (Investigations) | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA
Myocardial necrosis marker increased (Investigations) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 3 | NA | NA | NA | NA
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 2 | NA | NA | NA | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 2 | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Degenerative bone disease (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 2 | NA | NA | NA | NA
Tumour obstruction (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Demyelinating polyneuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Hepatic encephalopathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 2 | NA | NA | NA | NA
Acute kidney injury (Renal and urinary disorders) | 0 | 3 | 1 | 0 | 4 | NA | NA | NA | NA
Bladder tamponade (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Orchitis noninfective (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 3 | NA | NA | NA | NA
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 2 | NA | NA | NA | NA
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | NA | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | NA | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 0 | 2 | 0 | 2 | NA | NA | NA | NA
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_On- and Post-treatment (N=11) | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_On- and Post-treatment (N=46) | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel_On- and Post-treatment (N=49) | Arm 3: Gemcitabine/Nab-paclitaxel_On- and Post-treatment (N=45) | All Participants_On- and Post-treatment (N=151) | Run-in: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_Survival Period (N=0) | Arm 1: NIS793 + Spartalizumab + Gemcitabine/Nab-paclitaxel_Survival Period (N=0) | Arm 2: NIS793 + Gemcitabine/Nab-paclitaxel_Survival Period (N=0) | Arm 3: Gemcitabine/Nab-paclitaxel_Survival Period (N=0)
Anaemia (Blood and lymphatic system disorders) | 5 | 29 | 33 | 20 | 87 | NA | NA | NA | NA
Leukocytosis (Blood and lymphatic system disorders) | 1 | 3 | 0 | 2 | 6 | NA | NA | NA | NA
Leukopenia (Blood and lymphatic system disorders) | 1 | 4 | 2 | 3 | 10 | NA | NA | NA | NA
Neutropenia (Blood and lymphatic system disorders) | 5 | 11 | 9 | 9 | 34 | NA | NA | NA | NA
Neutrophilia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 7 | 4 | 4 | 17 | NA | NA | NA | NA
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 4 | NA | NA | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 | 4 | 9 | 4 | 18 | NA | NA | NA | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4 | 8 | 5 | 18 | NA | NA | NA | NA
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA
Constipation (Gastrointestinal disorders) | 1 | 16 | 16 | 12 | 45 | NA | NA | NA | NA
Diarrhoea (Gastrointestinal disorders) | 5 | 26 | 19 | 18 | 68 | NA | NA | NA | NA
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 4 | 3 | 8 | NA | NA | NA | NA
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 3 | NA | NA | NA | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 5 | 4 | 10 | NA | NA | NA | NA
Gingival bleeding (Gastrointestinal disorders) | 2 | 1 | 6 | 0 | 9 | NA | NA | NA | NA
Gingival hypertrophy (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Gingival swelling (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 2 | NA | NA | NA | NA
Haemorrhoids (Gastrointestinal disorders) | 1 | 1 | 3 | 0 | 5 | NA | NA | NA | NA
Ileal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Ileus (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | NA | NA | NA | NA
Nausea (Gastrointestinal disorders) | 7 | 20 | 27 | 20 | 74 | NA | NA | NA | NA
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 4 | 0 | 5 | NA | NA | NA | NA
Tongue coated (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Tongue disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Vomiting (Gastrointestinal disorders) | 3 | 10 | 18 | 12 | 43 | NA | NA | NA | NA
Asthenia (General disorders) | 5 | 12 | 16 | 11 | 44 | NA | NA | NA | NA
Chills (General disorders) | 1 | 3 | 2 | 5 | 11 | NA | NA | NA | NA
Fatigue (General disorders) | 7 | 23 | 18 | 14 | 62 | NA | NA | NA | NA
Mucosal inflammation (General disorders) | 1 | 5 | 4 | 1 | 11 | NA | NA | NA | NA
Oedema (General disorders) | 1 | 3 | 0 | 2 | 6 | NA | NA | NA | NA
Oedema peripheral (General disorders) | 4 | 11 | 15 | 8 | 38 | NA | NA | NA | NA
Pain (General disorders) | 1 | 2 | 1 | 1 | 5 | NA | NA | NA | NA
Pyrexia (General disorders) | 7 | 19 | 11 | 14 | 51 | NA | NA | NA | NA
Hepatobiliary disease (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
COVID-19 (Infections and infestations) | 1 | 13 | 6 | 5 | 25 | NA | NA | NA | NA
Infection (Infections and infestations) | 1 | 2 | 0 | 0 | 3 | NA | NA | NA | NA
Pneumonia (Infections and infestations) | 0 | 0 | 2 | 3 | 5 | NA | NA | NA | NA
Urinary tract infection (Infections and infestations) | 0 | 7 | 6 | 1 | 14 | NA | NA | NA | NA
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 4 | NA | NA | NA | NA
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 2 | 5 | NA | NA | NA | NA
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 2 | NA | NA | NA | NA
Alanine aminotransferase increased (Investigations) | 4 | 14 | 10 | 10 | 38 | NA | NA | NA | NA
Amylase increased (Investigations) | 1 | 5 | 2 | 2 | 10 | NA | NA | NA | NA
Aspartate aminotransferase increased (Investigations) | 4 | 13 | 9 | 7 | 33 | NA | NA | NA | NA
Blood alkaline phosphatase increased (Investigations) | 2 | 4 | 2 | 3 | 11 | NA | NA | NA | NA
Blood bilirubin increased (Investigations) | 0 | 1 | 5 | 4 | 10 | NA | NA | NA | NA
Blood creatinine increased (Investigations) | 0 | 3 | 1 | 0 | 4 | NA | NA | NA | NA
Blood lactate dehydrogenase increased (Investigations) | 0 | 2 | 3 | 1 | 6 | NA | NA | NA | NA
C-reactive protein increased (Investigations) | 0 | 4 | 2 | 0 | 6 | NA | NA | NA | NA
Gamma-glutamyltransferase increased (Investigations) | 4 | 1 | 1 | 2 | 8 | NA | NA | NA | NA
Lipase increased (Investigations) | 2 | 5 | 3 | 2 | 12 | NA | NA | NA | NA
Neutrophil count decreased (Investigations) | 2 | 7 | 8 | 9 | 26 | NA | NA | NA | NA
Platelet count decreased (Investigations) | 1 | 8 | 10 | 9 | 28 | NA | NA | NA | NA
Tri-iodothyronine decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Weight decreased (Investigations) | 2 | 2 | 6 | 5 | 15 | NA | NA | NA | NA
White blood cell count decreased (Investigations) | 0 | 3 | 3 | 3 | 9 | NA | NA | NA | NA
Decreased appetite (Metabolism and nutrition disorders) | 4 | 10 | 17 | 15 | 46 | NA | NA | NA | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 4 | 1 | 3 | 8 | NA | NA | NA | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 1 | 5 | NA | NA | NA | NA
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 8 | 6 | 9 | 24 | NA | NA | NA | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 4 | 2 | 3 | 10 | NA | NA | NA | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 2 | 6 | NA | NA | NA | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 9 | 7 | 2 | 21 | NA | NA | NA | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 4 | 5 | 8 | 18 | NA | NA | NA | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 5 | 2 | 14 | NA | NA | NA | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 1 | 4 | 8 | NA | NA | NA | NA
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 4 | NA | NA | NA | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 2 | 7 | NA | NA | NA | NA
Dizziness (Nervous system disorders) | 0 | 1 | 3 | 4 | 8 | NA | NA | NA | NA
Dysgeusia (Nervous system disorders) | 1 | 6 | 5 | 4 | 16 | NA | NA | NA | NA
Headache (Nervous system disorders) | 1 | 2 | 1 | 2 | 6 | NA | NA | NA | NA
Hypoaesthesia (Nervous system disorders) | 0 | 3 | 3 | 3 | 9 | NA | NA | NA | NA
Neuropathy peripheral (Nervous system disorders) | 0 | 5 | 11 | 5 | 21 | NA | NA | NA | NA
Neurotoxicity (Nervous system disorders) | 0 | 1 | 0 | 4 | 5 | NA | NA | NA | NA
Paraesthesia (Nervous system disorders) | 2 | 4 | 3 | 6 | 15 | NA | NA | NA | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 4 | 2 | 4 | 10 | NA | NA | NA | NA
Polyneuropathy (Nervous system disorders) | 1 | 5 | 5 | 1 | 12 | NA | NA | NA | NA
Anxiety (Psychiatric disorders) | 0 | 3 | 4 | 0 | 7 | NA | NA | NA | NA
Insomnia (Psychiatric disorders) | 1 | 4 | 3 | 7 | 15 | NA | NA | NA | NA
Haematuria (Renal and urinary disorders) | 0 | 3 | 1 | 0 | 4 | NA | NA | NA | NA
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 11 | 12 | 27 | NA | NA | NA | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 8 | 7 | 17 | NA | NA | NA | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 11 | 14 | 1 | 28 | NA | NA | NA | NA
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 1 | 4 | NA | NA | NA | NA
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3 | 1 | 9 | NA | NA | NA | NA
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 11 | 15 | 7 | 36 | NA | NA | NA | NA
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 3 | 3 | 1 | 7 | NA | NA | NA | NA
Erythema (Skin and subcutaneous tissue disorders) | 1 | 4 | 3 | 1 | 9 | NA | NA | NA | NA
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 3 | NA | NA | NA | NA
Onycholysis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 14 | 8 | 1 | 25 | NA | NA | NA | NA
Rash (Skin and subcutaneous tissue disorders) | 6 | 13 | 18 | 5 | 42 | NA | NA | NA | NA
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 10 | 1 | 0 | 13 | NA | NA | NA | NA
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 2 | 3 | 7 | NA | NA | NA | NA
Hypertension (Vascular disorders) | 1 | 3 | 4 | 2 | 10 | NA | NA | NA | NA
Hypotension (Vascular disorders) | 0 | 4 | 6 | 4 | 14 | NA | NA | NA | NA
Jugular vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA
Vein rupture (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | NA | NA | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. Novartis does not prohibit any investigator from publishing. Any publications from a single site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT04390763/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-11): https://cdn.clinicaltrials.gov/large-docs/63/NCT04390763/SAP_001.pdf